CLINICAL TRIAL: NCT03080025
Title: The Effects of a Cognitively-based Compassion Training on Health and Social Interaction in Depressed Patients and Their Partners
Brief Title: Social Interaction and Compassion in Depression
Acronym: SIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Emory University (Other); University of Arizona (Other); University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Beate Ditzen, Prof. Dr. phil. Dipl.- Psych. Beate Ditzen, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMP-CBC-247; Ethics Commission (Other: S-021/2016)
Record Dates: First submitted 2016-10-25; First posted 2017-03-15 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Depression; Couples (Persons)
Keywords: CBCT® (Cognitively Based Compassion-Training); Psychobiological Evaluation; Real Time Social Interaction; Eye-Tracking; Heart Rate Variability; IL-6; IL-1b; Cortisol; Alpha-Amylase; Randomised Controlled Trial; Compassion; Empathy; Relationship Quality; Interpersonal Relations; Stress
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBCT® for Couples (Experimental): The CBCT® (Cognitively Based Compassion-Training) for couples (CBCT®-fC) consists of a ten-week training program with a 2h group session weekly and daily home practice based on prerecorded guided mediations (Emory University, Atlanta, USA; Ozawa-de Silva & Negi, 2013). The ten weeks start with an overview and a take-home ideas for continuing practice. Furthermore the first and the 3rd module will be repeated once resulting in a total of ten weeks. Further couple- and dyadic exercises are added.
  It focuses on six essential key parts for the development of compassion:
  1. Developing attentional stability and clarity of the mind (Mindfulness)
  2. Cultivating insight into the nature of mental experience
  3. Cultivating self-compassion
  4. Developing impartiality
  5. Developing appreciation and affection for others
  6. Developing empathy and realizing engaged compassion
  Interventions: Behavioral: CBCT® (Cognitively Based Compassion-Training)
- Treatment as usual (TAU) (No Intervention): Treatment as usual: Primary care according to guidelines from the S3- and national healthcare guideline "Unipolar Depression" [S3-Leitlinie und Nationale VersorgungsLeitlinie (NVL) Unipolare Depression, Ärztliches Zentrum für Qualität in der Medizin], but excluding current psychotherapy after probatory session.

INTERVENTIONS:
Behavioral: CBCT® (Cognitively Based Compassion-Training) — The CBCT® (Cognitively Based Compassion-Training) as a secular approach was established as a structured protocol.
  The therapeutic tools are based on systemic approaches & techniques, which contains a resource- & solution orientation and the approach of Gottman's model of healthy relationships (e.g. trust and commitment - based on that - elements like "the positive perspective").
  Four dyadic exercises are introduced to enhance positive reciprocity between the romantic partners (based on concepts of couple communication training):
  a) Building mindful ability to talk, b) building mindful ability to listen (without reacting initially), c) appreciation in action - indulging the partner, d) "noticing, how the partner is doing something good for me" - gratefulness in action verbally/non-verbally. Finally, the "empathy exercise" has been added inspired by CBASP therapy for chronic major depression.
  Arms: CBCT® for Couples

SUMMARY:
The purpose of this study is to determine how a CBCT® (Cognitively Based Compassion-Training) for couples affect aspects of health and especially social interactions in depressed female patients and their romantic partners. compare healthy and depressed couples during an instructed positive real-time social interaction in the laboratory.

Furthermore the investigators aim to examine how social behavior and psychobiological indicators of health during real-time social interaction in the laboratory might be improved through CBCT® for couples.

DETAILED DESCRIPTION:
Objects:

Will a CBCT® (Cognitively Based Compassion-Training) for couples reduce the depressive symptomatic and the partners´ burden as well as improve behavioral, endocrine, physiological and immune responses during a real time social interaction in the laboratory.

Do couples with a depressed female partner differ from healthy control couples in behavioral, endocrine, physiological and immune responses during a instructed positive real-time social interaction in a laboratory setting?

ELIGIBILITY:
General inclusion criteria:

* being in a heterosexual relationship for two years or more
* agreement to participate in the study
* recurrent depression (ICD-10 F33.0 or F33.1, depressed females of the patient couples only)
* agreement of the patient couples to be randomized into the two treatment arms
* no mental disorders (healthy control group only)

General exclusion criteria:

* severe acute and chronic psychological ( suicidal tendency, acute affective bipolar disorders) or physical disorder (chronic diseases, severe diseases such as endocrinological, neurological, nephrological or hepatic disorders)
* being pregnant
* heavy smoking (more than 20 cigarettes daily) or alcohol abuse
* substance related abuse and addiction
* enrolling current couple therapy
* enrolling current individual therapy (except of probatory phase)
* enrolling current mindfulness or compassion based group training

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | 4 weeks after recruitment and 12 weeks after first test
  Change in depression score (observer rating Hamilton Depression Rating Scale [HDRS], self-rating Becks Depression Inventory [BDI]) after CBCT® (Cognitively Based Compassion Training) for couples in comparison to control TAU-group (treatment as usual).
Eye gaze patterns | 4 weeks after recruitment and 12 weeks after first test
  Changes in eye gaze patterns (total fixation time & fixation count) as behavioural component measured during standardised positive social interaction- pre & post training.
Circadian variation pattern of heart rate variability | 4 weeks after recruitment and 12 weeks after first test
  Changes in circadian variation pattern of heart rate variability pre & post training.

SECONDARY OUTCOMES:
Analysis of psychometrical self- and observer rating und their correlations | 4 weeks after recruitment and 12 weeks after first test
  Self- and observer ratings are:
  Berliner Social Support Skalen (BSSS) Compassionate Love Scale (CLS) Empathy Quotient (EQ) EuroQol five dimensions questionnaire (EQ5D) Evaluation of Social Systems (EVOS) UCLA-LS (HES) Inventory Interpersonal Probleme (IIP) Kentucky Inventory of Mindfulness Skills (KIMS) Partner Burden in Depression (PBD) Partnership Questionnaire (PFB) Patient Health Questionnaire (PHQ-9) Self Compassion Scale (SCS) Trier Inventar zum chronischen Stress (TICS)
Biopsychological concomitants of depressive disorders | 4 weeks after recruitment and 12 weeks after first test
  Saliva cortisol & alpha amylase, HbA1c, immune reactivity (Interleukin 1 beta [IL1b], Interleukin 6 [IL6], C-reactive protein [CRP]) and in epigenetical parameters (OXTR, SLC6A4) pre & post training.

CONTACTS AND LOCATIONS:
Overall Officials: Beate Ditzen, Prof. Dr., Principal Investigator — Institute of Medical Psychology, University Hospital Heidelberg
Locations (1):
- Institut of Medical Psychology at the Center for Psychosocial Medicine, University Hospital Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Winter F, Mander J, Jarczok MN, Warth M, Negi LT, Harrison T, Ditzen B, Aguilar-Raab C. Change Mechanism of Cognitively-Based Compassion Training for Couples with Depression: An Exploratory Empirical Investigation of Process Variables. J Integr Complement Med. 2022 Jul;28(7):591-599. doi: 10.1089/jicm.2022.0497. Epub 2022 May 17. PMID 35580123
- [Derived] Aguilar-Raab C, Jarczok MN, Warth M, Stoffel M, Winter F, Tieck M, Berg J, Negi LT, Harrison T, Pace TWW, Ditzen B. Enhancing Social Interaction in Depression (SIDE study): protocol of a randomised controlled trial on the effects of a Cognitively Based Compassion Training (CBCT) for couples. BMJ Open. 2018 Oct 4;8(9):e020448. doi: 10.1136/bmjopen-2017-020448. PMID 30287601